CLINICAL TRIAL: NCT05612178
Title: A Randomized Placebo-controlled Study to Evaluate the Safety and Effects of Repeated Doses of 3BNC117-LS and 10-1074-LS on Persistent Viral Reservoirs in People Living With HIV and on Suppressive Antiretroviral Therapy
Brief Title: A Study to Evaluate the Safety and Effects of Repeated Doses of 3BNC117-LS and 10-1074-LS on Persistent Viral Reservoirs in People Living With HIV and on Suppressive Antiretroviral Therapy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10001037; 001037-I
Record Dates: First submitted 2022-11-09; First posted 2022-11-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01-16

CONDITIONS: HIV-1
Keywords: bNAb; HIV Reservoir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 3BNC117-LS and 10-1074-LS (Experimental): Participants will receive three intravenous infusions of 3BNC117-LS (dosed at 30 mg /kg) and 10-1074-LS (dosed at 10 mg/kg) at weeks 0, 20 and 40.
  Interventions: Biological: 3BNC117-LS; Biological: 10-1074-LS
- Placebo (Placebo Comparator): Participants will receive three intravenous infusions of placebo (Sterile Saline) at weeks 0, 20 and 40.
  Interventions: Other: Sterile Saline

INTERVENTIONS:
Biological: 3BNC117-LS — Participants will receive three intravenous infusions of 3BNC117-LS (dosed at 30 mg /kg) and 10-1074-LS (dosed at 10 mg/kg) or placebo at weeks 0, 20 and 40.
  Arms: 3BNC117-LS and 10-1074-LS
Biological: 10-1074-LS — Participants will receive three intravenous infusions of 3BNC117-LS (dosed at 30 mg /kg) and 10- 1074-LS (dosed at 10 mg/kg) or placebo at weeks 0, 20 and 40.
  Arms: 3BNC117-LS and 10-1074-LS
Other: Sterile Saline — Participants will receive three intravenous infusions of 3BNC117-LS (dosed at 30 mg /kg) and 10-1074-LS (dosed at 10 mg/kg) or placebo at weeks, 20 and 40.
  Arms: Placebo

SUMMARY:
Background:

Antiretroviral therapy (ART) can suppress HIV to undetectable levels in people, but the virus rebounds quickly if the drug treatment is stopped; this is because HIV can remain dormant in a pool of blood cells called the persistent viral reservoir (PVR). Yet lifelong ART is expensive and can lead to serious side effects over the long term. Some drugs may be more effective at reducing the PVR.

Objective:

To see if 2 study drugs (3BNC117-LS and 10-1074-LS) are safe and if they can lower the number of HIV-infected blood cells in people with HIV who are on ART.

Eligibility:

People aged 18 to 70 years with HIV who are on ART.

Design:

Participants will be screened. They will have a physical exam and blood and urine tests. They will undergo leukapheresis. Leukapheresis is a procedure where blood is drawn from a needle in one arm. The blood will pass through a machine that separates out the white blood cells. The remaining blood will be given back through a second needle in the other arm.

The study drugs or placebo (normal saline) will be administered 3 times at 20-week intervals. The drugs will be given through a tube attached to a needle inserted into a vein in the arm. This will take 1 hour. Some participants will receive only a saline solution. They will not know if they are getting the drugs or the placebo.

Participants will undergo leukapheresis up to 4 more times during the study.

Participants will have follow-up visits every 10 weeks until the study ends.

DETAILED DESCRIPTION:
Study Description:

This is randomized placebo-controlled study of the safety and virologic activity of the 3BNC117-LS plus 10-1074-LS broadly neutralizing antibody (bNAb) combination during standard antiretroviral therapy (ART).

Participants will be enrolled sequentially and randomized to receive 3BNC117-LS plus 10-1074-LS or placebo (sterile saline) at a 1:1 ratio. Participants will receive two intravenous infusions of 3BNC117-LS (dosed at 30 mg/kg) and 10-1074-LS (dosed at 10 mg/kg) or placebo at weeks 0 and 20. Participants will remain on ART during the study.

Objectives:

Primary Objectives:

-To evaluate the safety and tolerability of repeated doses of 3BNC117-LS and 10-1074-LS in adults living with human immunodeficiency virus (HIV) during suppressive ART.

Secondary Objectives:

* To evaluate the impact of 3BNC117-LS and 10-1074-LS on intact human immunodeficiency type 1 (HIV-1) proviruses over time in adults living with HIV during suppressive ART.
* To determine the effects of repeated doses of 3BNC117-LS and 10- 1074-LS during suppressive ART on HIV-1 specific cellular immune responses by enzyme-linked immunosorbent spot (ELISpot).
* To describe the pharmacokinetic parameters of the repeated doses of 3BNC117-LS and 10-1074-LS in adults living with HIV during suppressive ART.

Exploratory Objectives:

* To characterize the HIV-1 reservoir in peripheral blood during and following repeated doses of 3BNC117-LS and 10-1074-LS during suppressive ART.
* To evaluate effects on HIV-1 transcriptional activity during and following repeated doses of 3BNC117-LS and 10-1074-LS during suppressive ART.
* To characterize host HIV-1 specific humoral, cellular and innate immune responses during and following repeated doses of 3BNC117-LS and 10-1074-LS during suppressive ART.
* To correlate HIV-1 specific immune responses and effects on intact proviruses.
* To correlate virologic outcomes with bNAb sensitivity of reservoir proviruses.

Endpoints:<TAB>

Primary Endpoints:

-The occurrence of solicited and unsolicited grade 3 or higher adverse events (AE) (including confirmed laboratory abnormalities) that are possibly, probably, or definitely related to 3BNC117-LS and/or 10- 1074-LS, or premature study treatment discontinuation due to an AE (regardless of grade).

Secondary Endpoints:

* The occurrence of serious adverse events, regardless of relationship to 3BNC117-LS and/or 10-1074-LS.
* Change in the intact proviral reservoir size, measured by quadruplex polymerase chain reaction (Q4PCR) and/or intact proviral deoxyribonucleic acid assay (IPDA), from baseline to weeks 40 and

  80 after dosing with 3BNC117-LS and 10-1074-LS during suppressive ART.
* Changes in HIV-1 specific T cell immune responses in peripheral blood, measured by ELISpot, before, during and after dosing with 3BNC117-LS and 10-1074-LS during suppressive ART.
* Pharmacokinetic parameters (including: peak concentrations, half- life, area under curve and clearance rate) of repeated doses of 3BNC117-LS and 10-1074-LS during suppressive ART.

Exploratory Endpoints:

* Size of the latent HIV-1 reservoir, measured by quantitative viral outgrowth assay (QVOA) and/or other appropriate assays, before, during and after dosing with 3BNC117-LS and 10-1074-LS during suppressive ART.
* Composition of the intact proviral reservoir before and after immunotherapy with 3BNC117-LS and 10-1074-LS during suppressive ART by Q4PCR or other appropriate assays that may become available.
* The half-life of the HIV-1 intact proviral reservoir during 3BNC117- LS and 10-1074-LS therapy and ART suppression.
* HIV-1 transcriptional activity as determined by spliced and unspliced HIV-1 ribonucleic acid (RNA) in circulating total CD4+ T cells and/or other appropriate assays, before, during and after dosing with 3BNC117-LS and 10-1074-LS during suppressive ART.
* Changes in HIV-1 specific T cell immune responses in peripheral blood, measured by assays such as polyfunctional intracellular cytokine staining (ICS) and viral inhibition assay before, during and after immunotherapy with 3BNC117-LS and 10-1074-LS during suppressive ART.
* Changes in antibody dependent cell-mediated cytotoxicity (ADCC) against HIV-1-infected CD4+ T-cells by ex vivo autologous natural killer cells before and after immunotherapy with 3BNC117-LS and 10-1074-LS during suppressive ART.
* Correlation between magnitude, breadth and functionality of HIV-1 specific T cell immune responses and effects on intact proviruses.
* Correlation between changes in intact proviruses and bNAb sensitivity of reservoir proviruses determined by Env sequencing.
* Correlation between HIV-1 transcriptional activity and changes in the composition of the intact proviral reservoir.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Ability to provide informed consent;
2. Stated willingness to comply with all study procedures and availability for the duration of the study;
3. Adult persons of any sex or gender, aged 18 years to 70;
4. Confirmed HIV-1 infection and clinically stable;
5. On antiretroviral therapy with plasma HIV-1 RNA levels of < 50 copies/mL and no reported interruption of ART for 7 consecutive days or longer for at least 96 weeks. NOTE: At least two viral load (VL) measurements within 48 weeks prior to the screening visit must be available for review. A single plasma HIV-1 RNA > 50 copies/mL but < 200 copies/mL over 48 weeks that is followed by an HIV-1 RNA < 50 copies/mL is permitted;
6. Current CD4+ T cell counts > 300 cells/mcL;
7. For participants who can become pregnant (i.e., participants who have not been postmenopausal for at least 24 consecutive months, who have had menses within the preceding 24 months, or who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy), must have a negative pregnancy test at screening and within 48 hours prior to day 0; NOTE: Participant-reported history is acceptable as documentation of hysterectomy and bilateral oophorectomy, tubal ligation, tubal micro-inserts, and vasectomy.
8. Participants who can become pregnant must agree to use adequate measures to prevent pregnancy. This includes the use an effective method of contraception for the study duration. Contraception must be used from 10 days prior to the first dose of the investigational products (IPs), while receiving the IPs and during study follow up. Acceptable methods of contraception include:

   * Contraceptive subdermal implant
   * Intrauterine device or intrauterine system
   * Combined estrogen and progestogen oral contraceptive
   * Injectable progestogen
   * Contraceptive vaginal ring
   * Percutaneous contraceptive patches

   NOTE: Partner sterilization with documentation of azoospermia prior to the participant's entry into the study, and this partner is the sole partner for that participant, will be allowed. The documentation of partner sterility can come from the site personnel s review of medical records, medical examination and/or semen analysis, or medical history interview provided by the participant or the partner. Self-reported documentation of reproductive potential should be entered in the source documents.
9. Participants who can impregnate a partner and who are engaging in sexual activity that could lead to pregnancy must agree to use condoms from 10 days prior to the first dose of the IPs, while receiving the IPs and during study follow up to avoid impregnating a partner who can get pregnant.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. History of AIDS-defining illness within 3 years prior to enrollment;
2. History of systemic corticosteroids (e.g., an equivalent dose of prednisone of > 20 mg daily for >14 days), immunosuppressive anti-cancer, interleukins, systemic interferons, systemic chemotherapy or other medications considered significant by the trial physician within the last 6 months;
3. Any clinically significant acute or chronic medical condition (e.g. such as autoimmune diseases, cirrhosis, active malignancy that may require systemic chemotherapy or radiation therapy), other than HIV infection, that in the opinion of the investigator would preclude participation;
4. Hepatitis B or C infection as indicated by the presence of Hepatitis B surface antigen (HBsAg) or hepatitis C virus RNA (HCV-RNA) in blood. NOTE: Participants with a positive test for HCV antibody and a negative test for HCV RNA are eligible;
5. Participants with known hypersensitivity to any constituent of the investigational products;
6. Pregnancy or lactation;
7. ART initiated during acute infection (defined as p24, HIV nucleic acid amplification technique [NAAT], or HIV RNA PCR positive, and negative or indeterminate HIV antibody testing);
8. Laboratory abnormalities in the parameters listed below:

   * Absolute neutrophil count < 1,000 cells/microliter
   * Hemoglobin < 10 gm/dL
   * Platelet count < 100,000 cells/microliter
   * ALT > 1.5 x ULN
   * AST > 1.5 x ULN
   * Total bilirubin > 1.5 x ULN
   * Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m^2
9. Any history of receipt of HIV-1 mAb therapy or HIV vaccine;
10. Participation in any clinical study of an investigational product within 12 weeks prior to study entry (day 0) or expected participation in such a study during this study;
11. Any approved or experimental non-HIV vaccination (e.g., SARS-CoV-2, hepatitis B, influenza, pneumococcal polysaccharide) received within 2 weeks prior to study enrollment (day 0);
12. Inability to undergo leukapheresis due to poor venous access or other medical conditions;
13. Active drug or alcohol use or any other pattern of behavior that, in the opinion of the investigator, would interfere with adherence to study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Solicited and unsolicited grade 3 or higher adverse events | Week 0 to End of Study
  The occurrence of solicited and unsolicited grade 3 or higher adverse events (AE) (including confirmed laboratory abnormalities) that are possibly, probably, or definitely related to 3BNC117-LS and/or 10-1074-LS, or premature study treatment discontinuation due to an AE (regardless of grade).

SECONDARY OUTCOMES:
Occurrence of Serious Adverse Events | Week 0 to End of Study
  The occurrence of serious adverse events, regardless of relationship to 3BNC117-LS and/or 10-1074-LS.
Change in the intact proviral reservoir size | Baseline to Weeks 40 and 80
  Change in the intact proviral reservoir size, measured by Q4PCR and /or IPDA, from baseline to weeks 40 and 80 after dosing with 3BNC117-LS and 10-1074-LS during
Changes in HIV-1 specific T cell immune responses in peripheral blood | Throughout
  Changes in HIV-1 specific T cell immune responses in peripheral blood, measured by ELISpot, before, during and after dosing with 3BNC117 LS and 10-1074-LS during suppressive ART.
Pharmacokinetic parameters | Throughout
  Pharmacokinetic parameters (including: peak concentrations, halflife, area under curve and clearance rate) of repeated doses of 3BNC117-LS and 10-1074-LS during suppressive ART.

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Sneller, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - The Rockefeller University, New York, New York

REFERENCES:
- [Background] Mendoza P, Gruell H, Nogueira L, Pai JA, Butler AL, Millard K, Lehmann C, Suarez I, Oliveira TY, Lorenzi JCC, Cohen YZ, Wyen C, Kummerle T, Karagounis T, Lu CL, Handl L, Unson-O'Brien C, Patel R, Ruping C, Schlotz M, Witmer-Pack M, Shimeliovich I, Kremer G, Thomas E, Seaton KE, Horowitz J, West AP Jr, Bjorkman PJ, Tomaras GD, Gulick RM, Pfeifer N, Fatkenheuer G, Seaman MS, Klein F, Caskey M, Nussenzweig MC. Combination therapy with anti-HIV-1 antibodies maintains viral suppression. Nature. 2018 Sep;561(7724):479-484. doi: 10.1038/s41586-018-0531-2. Epub 2018 Sep 26. PMID 30258136
- [Background] Niessl J, Baxter AE, Mendoza P, Jankovic M, Cohen YZ, Butler AL, Lu CL, Dube M, Shimeliovich I, Gruell H, Klein F, Caskey M, Nussenzweig MC, Kaufmann DE. Combination anti-HIV-1 antibody therapy is associated with increased virus-specific T cell immunity. Nat Med. 2020 Feb;26(2):222-227. doi: 10.1038/s41591-019-0747-1. Epub 2020 Feb 3. PMID 32015556
- [Background] Gaebler C, Nogueira L, Stoffel E, Oliveira TY, Breton G, Millard KG, Turroja M, Butler A, Ramos V, Seaman MS, Reeves JD, Petroupoulos CJ, Shimeliovich I, Gazumyan A, Jiang CS, Jilg N, Scheid JF, Gandhi R, Walker BD, Sneller MC, Fauci A, Chun TW, Caskey M, Nussenzweig MC. Prolonged viral suppression with anti-HIV-1 antibody therapy. Nature. 2022 Jun;606(7913):368-374. doi: 10.1038/s41586-022-04597-1. Epub 2022 Apr 13. PMID 35418681
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001037-I.html